CLINICAL TRIAL: NCT00112333
Title: Defining Central Circuits of Visceral Pain
Brief Title: Defining Central Circuits of Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Braden Kuo, MD, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2003-P-001304
Record Dates: First submitted 2005-06-01; First posted 2005-06-02 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Dyspepsia
Keywords: Dyspepsia, fMRI
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: fMRI — A liquid meal (Ensure 1Kcal/cc) will be infused into the stomach via a nasogastric tube at a rate of 60cc/min till the subject reaches maximal satiety. The amount of liquid meal will differ per subject.

SUMMARY:
The purpose of the study is to use functional Magnetic Resonance Imaging (MRI) to help us understand what parts of the subject's brain are involved when he experiences visceral pain, or pain in the gut. To stimulate the brain, he will be infused with a liquid meal (Ensure) into his stomach until he is maximally full. Magnetic resonance imaging (MRI) is a technique for making images (pictures) of the brain; it uses magnetic fields and radio waves and is not harmful. This study uses a new investigational technique called functional MRI (fMRI), which is a very fast MRI technique that will allow the investigators to evaluate changes in how blood flows to parts of his brain.

DETAILED DESCRIPTION:
Dyspepsia, a condition characterized by upper abdominal discomfort, is one of the most common types of pains in clinical practice and is one of the most common reasons for visits to primary care physicians and gastroenterologists. But relative to somatic pain, little fundamental information is known about visceral pain syndromes such as dyspepsia and irritable bowel syndrome. Recent exciting advances in neuroimaging such as functional magnetic resonance imaging (fMRI) have allowed investigators to interrogate neural signal changes in humans in a wide variety of pain conditions. But to date neuroimaging has not provided details of activation in specific neural circuits that are important in visceral pain. In these experiments we will focus on specific regions of interest (ROI's) that have shown to be relevant in animal models of pain circuitry including the dorsal column nuclei, the thalamus, the hypothalamus, the amygdala and the periaqueductal gray.

The specific aims of our proposed project are:

1. To measure fMRI signal in primary visceral afferent pain pathways (dorsal column nuclei and thalamus) in normal human subjects and in patients with dyspepsia following instilling a liquid meal at a fixed rate into the stomach until maximal satiety, a surrogate model of dyspepsia.
2. To measure fMRI signal in autonomic pathways (hypothalamus and amygdala) and in endogenous analgesic pathways (periaqueductal gray/PAG) in normal human subjects and in patients with dyspepsia using the above model.
3. To correlate physiological parameters (heart rate, skin conductance, respiratory rate) to hedonic ratings (ratings on a visual analogue scale of satiety, nausea, bloating, and pain) during the liquid meal stimulus in normal human subjects and patients with dyspepsia.

In all these experiments we will correlate alterations in psychophysical measures which have traditional measures of pain response (e.g., pain and other hedonic ratings, physiological monitoring such as heart rate, etc) with the changes in fMRI signal in specific areas of the brain.

ELIGIBILITY:
Inclusion Criteria:

* Right handed men and non-pregnant women ages 18 to 64

Exclusion Criteria:

* Diabetes
* History of aspiration or severe respiratory complications linked to gastrointestinal disease
* Use of any over the counter medications within 7 days of the study
* Current or previous history of gastric surgery
* Use of any medications which may alter gastrointestinal motility

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2003-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Dyspepsia | after session

SECONDARY OUTCOMES:
Meal fullness | after session

CONTACTS AND LOCATIONS:
Overall Officials: Braden Kuo, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Martinos Center for Biomedical Imaging, Charlestown, Massachusetts, United States